CLINICAL TRIAL: NCT03891745
Title: Emergence From Prone or Supine Extubation After Lomber Spinal Surgery
Brief Title: Prone or Supine Extubation in Lomber Spinal Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: 2018-0117
Record Dates: First submitted 2019-03-04; First posted 2019-03-27 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prone group: prone extubation
- supine group: supine extubation

SUMMARY:
The aim of this study was to investigate the emergence quality of patients extubated on prone or supine position after lumbar spinal surgery.

60 patients with ASA I-II who underwent lumbar spinal surgery between 18-65 years of age were included in the study. Patients with difficult intubation, BMI> 35kg / m2, asthma and reactive airway problems, cardiovascular disease and obstructive sleep apnea will not be included in the study. Initial data will be recorded after standard monitorization. Induction is made by 2 mg / kg propofol, 1 mg / kg fentanyl and 0.5 mg / kg rocuronium will be added for muscle relaxation. Patients with adequate muscle relaxation will be intubated with appropriate endotracheal tube and mechanical ventilation will be initiated. Patients who are then given prone positions on the operating table will be supported with side gels. The head will be placed in the face gel in a neutral position. For intraoperative analgesia, remifentanil infusion at 0.2mcg / kg / min will be applied.

After laminectomy is completed and control of bleeding, 1 mg / kg Tramalol and 2 mg / kg Metaclopromide will be applied to all patients. At the end of the skin stitching, the inhalation agent will be closed and the fresh gas will be turned 6 lt 100% O2. Patients who want to be extubated in the prone position are left in this position while the other patients will be placed on the stretcher in a supine position for a short time. Patients will be decurarized be neostigmin with atropine. Extubation will be performed in both positions when spontanous ventilation begins at a tidal volume of 6ml / kg and a frequency of 12-20 / min. All the measures will be taken to ensure airway safety while the patient is extubated pron. The stretcher will be brought to the side of the operating table, investigator will be ready for reintubation and all the necessary persons will be with the patient. Aspiration frequency will be recorded for each patient. During recovery after extubation, the severity of cough will be evaluated as mild (only once), less (more than one but not continuous) and severe (continuously for 5 seconds). Aldrate scores of patient will be recorded and first 9-10 time is estimated from extubation time. Vomiting, nausea, respiratory insufficiency, inability to control the airway and obvious desaturation if seen are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 18-65 years old
* need spinal surgery

Exclusion Criteria:

* difficult intubation
* BMI> 35kg / m2
* asthma and reactive airway problems
* cardiovascular disease
* obstructive sleep apnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lomber spinal surgery will be sected
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Modified-Aldrete Scale | 1 hour
  Modified-Aldrete Scale: It is used for postanesthesia recovery status. Its range from 0-10. When the values is between 9-10, the patient is ready to transport from postanesthetic care unit.
Ricker's Agitation Scale | 1 hour
  Ricker's Agitation Scale: This scale is used for sedation agitation status of the patients under sedatives in intensive care units or postanesthetic care units. Its range is between 1-7. The optimum wanted values are 3-4.

CONTACTS AND LOCATIONS:
Locations (1):
- Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No